CLINICAL TRIAL: NCT05241938
Title: Computer-guided Selective Laser Trabeculoplasty (PSLT) in the Treatment of Ocular Hypertension and Open-angle Glaucoma Compared to Prostaglandin Analogue Eye Drops: a Non-inferiority Randomized Clinical Trial
Brief Title: PSLT Compared to Prostaglandin Analogue Eye Drops
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Helena Messinger Pakter, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44489320.7.0000.5327
Record Dates: First submitted 2022-01-27; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pattern Selective Laser Trabeculoplasty (Experimental): PSLT will be performed using the Pascal Streamline 577 laser (Topcon Inc., Tokyo, Japan). The laser spot is directed at the anterior chamber angle encompassing the pigmented and non-pigmented trabecular meshwork. Laser power is titrated by placing a laser mark in the lower quadrant with an exposure duration of 10 milliseconds (ms). The initial energy of 500 megawatts (mW) is selected and the power is reduced or increased until a slight whitening of the trabecular meshwork is minimally noticed. This power is then maintained and the pulse duration is automatically reduced to 5ms to produce invisible injury. The treatment is administered in 32 steps, each pattern consists of 36 stitches: 3 rows of 13 stitches each (total of 1152), with zero space between adjacent stitches.
  Interventions: Procedure: PSLT
- Prostaglandin analogue eye drops (Active Comparator): Prostaglandin analogue eye drops (latanoprost, bimatoprost or travoprost) will be prescribed
  Interventions: Drug: Prostaglandin analogue eye drops

INTERVENTIONS:
Procedure: PSLT — PSLT will be performed under topical anesthesia (proxymetacaine hydrochloride 5mg/ml eye drops) using a mirrored gonioscopy lens (Latina Ocular Instruments). A α2 agonist hypotensive eye drops (0.2% brimonidine tartrate) and 2% pilocarpine eye drops are applied 40 minutes before the procedure. After laser treatment, the patient will be instructed to use non-steroidal anti-inflammatory eye drops (thrice daily for 7 days).
  Other Names: Pattern Selective Laser Trabeculoplasty
  Arms: Pattern Selective Laser Trabeculoplasty
Drug: Prostaglandin analogue eye drops — Prostaglandin analogue eye drops will be prescribed to be used continuously once a day in the fellow eye.
  Other Names: Topical treatment
  Arms: Prostaglandin analogue eye drops

SUMMARY:
This study aims to compare the efficacy of PSLT and the topical use of prostaglandin-like hypotensive eye drops in the treatment of ocular hypertensive or glaucomatous patients in decreasing intraocular pressure and measuring changes in functional, structural and biomechanical parameters evaluated by computerized perimetry and optical coherence tomography (OCT) related to pressure change resulting from treatments

DETAILED DESCRIPTION:
Patients with a diagnosis of ocular hypertension or bilateral glaucoma, naive or on treatment with up to two classes of hypotensive eye drops will be invited to participate in the study.

These patients will have both eyes included in the study. A randomization will be made to allocate one eye to receive treatment with PSLT (treatment group), while the contralateral eye will receive treatment with prostaglandin eye drops (control).

Patients will be followed up for 12 months and periodically tonometry, computerized perimetry, water overload test and OCT will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension (IOP ≥ 24 mmHg in both eyes) or diagnosis of open-angle glaucoma (POAG) in both eyes
* Proper visualization of angle structures and 360 degree open angles in both eyes
* No previous intraocular surgery with the exception of phacoemulsification with intraocular lens implantation
* No use of systemic medications known to increase IOP

Exclusion Criteria:

* Patients using more than two glaucoma medications
* Evidence of any other eye disease that could affect IOP measurement
* Diagnosis of other types of glaucoma
* Patient with mean deviation (MD) less than -12 decibels (dB) on visual perimetry (severe disease)
* Patients with unilateral glaucoma

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure change | 1 week, 2 months, 9 months, 12 months
  Intra-ocular pressure change will be similar in both groups

SECONDARY OUTCOMES:
Structural damage | 1 week, 9 months, 12 months
  Changes in nerve fiber layer and ganglion cell layer thickness as measured by OCT will be assessed
Functional damage | 1 week, 9 months, 12 months
  Changes in visual function as measured by computerized perimetry will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Helena Pakter, MD. PhD, Principal Investigator — UFGRS
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No